CLINICAL TRIAL: NCT00325624
Title: Diabetes Risk Evaluation and Management Tele-monitoring Study (DREAM-Tel)
Acronym: DREAM-Tel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Battlefords Tribal Council Indian Health Services (Unknown); SaskTel (Industry)
Responsible Party: Principal Investigator, Sheldon Tobe, Associate Professor of Medicine, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 2006-04
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Hypertension; Diabetes Mellitus
Keywords: Blood Pressure; Diabetes mellitus; Hypertension; Home Care; Glucometer
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

INTERVENTIONS:
Device: Bluetooth-enabled Glucometer — blood glucose information provided to health care providers

SUMMARY:
The purpose behind the proposed research is that diabetes care in First Nations people can be improved by involvement of a Home Care team providing diabetes education and management, supported by emerging technology, specifically Bluetooth-enabled glucometers and blood pressure monitors, capable of transmitting their data to a web environment in tabulated and graphical format available for remote viewing.

DETAILED DESCRIPTION:
Diabetes mellitus is a systemic disease that produces a diverse array of complications. The pathogenesis of these complications refers back to two factors, one of which (high blood glucose) alters proteins leading to tissue and blood vessel damage, while the other (high blood pressure), exacerbates the vascular damage causing further damage to target organs. Our long term goal is to achieve targets for blood glucose and blood pressure as outlined by Clinical Practice Guidelines.

Despite current Clinical Practice Guidelines and evidence-based practice by the medical community, including family physicians and the Home Care team, blood glucose control in general and in the First Nations community specifically is not meeting targets. Poor control of blood glucose in type 2 diabetes dramatically increases the risk of heart disease, stroke, vascular limb loss, blindness, kidney disease and the need for dialysis. Control of blood glucose levels prevents these complications. Additionally, the intensification of diabetes control, including the initiation of insulin, is not easily done during a regular primary care visit. The lack of intensification of diabetes management in people with poorly controlled diabetes has been referred to as 'clinical inertia'. While subjects referred to specialists have somewhat better control of diabetes, more than 50% still failed to have intensification of diabetes management within four months of a lab report showing a high level of A1c. Multidisciplinary care can overcome clinical inertia, even in difficult practice settings. Finally, the emerging technology of Bluetooth-enabled devices and secure web-based monitoring logs allows health care providers for the first time to remotely monitor progress providing a higher level of confidence in self blood glucose monitoring (SBGM) and blood pressure results. Based on these facts, the experimental focus of this proposal is on the introduction of a Home Care Team diabetes management program that can provide intensification of diabetes management right in the patient's home, supported by the emerging technology of Bluetooth- enabled devices. The specific aims are designed to provide a comprehensive assessment of the impact of the introduction of this program.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes with baseline A1c > 8.0 % on diet or medical therapy with no history of diabetic ketoacidosis.
* Patients must be greater than or equal to 18 years of age.
* Written informed consent must be obtained prior to admission to this study.

Exclusion Criteria:

* Hypoglycemic therapy and A1c<8.0%
* New York Heart Association Stage III-IV congestive heart failure. This will eliminate approximately 2% of people with diabetes based on the Strong Heart Study Data.
* Suspected secondary hypertension due to any cause (e.g. pheochromocytoma,coarction of the aorta or renal insufficiency.)
* Unstable angina, myocardial infarction, or revascularization within the last 3 months.
* Angioedema.
* Cerebrovascular event, including stroke or transient ischemic attack, within the last six months.
* Creatinine >250 umol/L
* Cerebral Vascular event, including strike or transient ischemic attack, within the last six months.
* Connective tissue disorders (e.g.lupus, rheumatoid arthritis)
* Active hepatic disease as indicated by AST and ALT >2X the upper limit of normal; serum bilirubin >1.5X upper limit of normal, or serum albumin <3.0 gm/dl.
* Severe systemic or malignant disease(which could reasonably be expected to be fatal or life-threatening during the course of the study.)
* Pregnancy. It is expected that some women will want to exit the study to become pregnant (5% of female enrollees).
* Factors suggesting low likelihood of compliance with the protocol (e.g current alcohol abuse, history of unreliability in keeping appointments or taking medications.
* Any medical condition that study physicians believe would interfere with study participation or evaluation of results.
* Mental incapacity and/or cognitive impairment on the part of the patient that would preclude adequate understanding of, or cooperation with, the study protocol.
* Participation in any clinical trial of any investigational medication within 3 months prior to this trial. This is unlikely because clinical trials among First Nations people are rare.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
A1c | 1 year
  Change of A1c over 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon W Tobe, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; George Pylypchuk, MD, FRCP(C), Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Battleford Tribal Council Indian Health Services, North Battleford, Saskatchewan

REFERENCES:
- [Derived] Tobe SW, Wentworth J, Ironstand L, Hartman S, Hoppe J, Whiting J, Kennedy J, McAllister C, Kiss A, Perkins N, Vincent L, Pylypchuk G, Lewanczuk RZ. DreamTel; Diabetes risk evaluation and management tele-monitoring study protocol. BMC Endocr Disord. 2009 May 9;9:13. doi: 10.1186/1472-6823-9-13. PMID 19426530